CLINICAL TRIAL: NCT04721431
Title: The Affect of Obesity to Muscle Tone and Viscoelastic Properties
Brief Title: The Investigation of Mechanical Properties in Obesity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Assistant of professeur, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020/101
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Body Fat Disorder; Obesity; Muscular Tone; Viscoelasticity
Keywords: Body mass index; Tone; Viscoelasticity; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The people will assigned to groups depend on body mass index. The biceps brachii (BB), biceps femoris (BF) tone, and viscoelastic properties (stiffness and elasticity) will be evaluated bilaterally using the ''MyotonPRO'' device.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal (Experimental): Body mass index must to be in range limits (18.5-24.9 kg/meter square)
  Interventions: Diagnostic Test: Myotonometric assessment
- Overweight (Experimental): Body mass index must to be in range limits (25-29.9 kg/meter square)
  Interventions: Diagnostic Test: Myotonometric assessment
- Obese (Experimental): Body mass index must to be in range limits (30-34.9 kg/meter square)
  Interventions: Diagnostic Test: Myotonometric assessment

INTERVENTIONS:
Diagnostic Test: Myotonometric assessment — MyotonPro device is vertically placed on the muscle, a probe (3 mm diameter) creates constant pre-excitations (0.18 N) and generates short-term (15 ms), low-force (0.4 N) mechanical stimulations.These stimulations induce damped natural oscillations in the tissue and the device records these oscillations using an accelerometer. Muscle tone, elasticity, and stiffness are calculated separately by the device

SUMMARY:
The study will demonstrate the relation between muscle tone and viscoelastic properties with the body mass index.

DETAILED DESCRIPTION:
Obesity is an increasingly important health problem. It can be defined as excessive fat accumulation. Obesity is a low-severity systemic inflammatory condition that predisposes to chronic diseases.Obesity is closely related to adipose tissue, it can have direct or indirect effects on physical activity and musculoskeletal system. The systems working with oscillation techniques, subcutaneous tissue thickness may affect the probe stroke of the device and oscillation in the tissue. In previous studies were investigated mechanical properties, and BMI used as exclusion criteria is over 30 kg/meter square or keeping it at certain intervals (18-28 kg /meter square) but this proof is not demonstrated and still lack.This study is planned to determine the relation of mechanical properties (tone, stiffness and elasticity) obtained by myotonometric assessment with body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (range; 18 - 35 kg/meter square)

Exclusion Criteria:

* Had any systemic or metabolic disease, psychological illness, or drug use,
* Had any disease that may cause muscle disease or muscle atrophy,
* musculoskeletal surgery for the last 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Stiffness obtained from myotonometric assessment | Baseline
  Myoton device stimulations create natural oscillations in the tissue and records these oscillations using an accelerometer. Stiffness (N/m) is calculated by device
Tone obtained from myotonometric assessment | Baseline
  Myoton device stimulations create natural oscillations in the tissue and records these oscillations using an accelerometer. Tone (Hz) is calculated by device
Elasticity obtained from myotonometric assessment | Baseline
  Myoton device stimulations create natural oscillations in the tissue and records these oscillations using an accelerometer. Elasticity (log) is calculated by device.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Usgu, Principal Investigator — hku
Locations (1):
- Hasan kalyoncu üniversity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mechelli F, Arendt-Nielsen L, Stokes M, Agyapong-Badu S. Validity of Ultrasound Imaging Versus Magnetic Resonance Imaging for Measuring Anterior Thigh Muscle, Subcutaneous Fat, and Fascia Thickness. Methods Protoc. 2019 Jul 10;2(3):58. doi: 10.3390/mps2030058. PMID 31295936
- [Background] Wood S, Pearsall DJ, Ross R, Reid JG. Trunk muscle parameters determined from MRI for lean to obese males. Clin Biomech (Bristol). 1996 Apr;11(3):139-144. doi: 10.1016/0268-0033(95)00018-6. PMID 11415611
- [Background] Tas S, Yilmaz S, Onur MR, Soylu AR, Altuntas O, Korkusuz F. Patellar tendon mechanical properties change with gender, body mass index and quadriceps femoris muscle strength. Acta Orthop Traumatol Turc. 2017 Jan;51(1):54-59. doi: 10.1016/j.aott.2016.12.003. Epub 2016 Dec 20. PMID 28010997
- [Result] Kocur P, Tomczak M, Wiernicka M, Goliwas M, Lewandowski J, Lochynski D. Relationship between age, BMI, head posture and superficial neck muscle stiffness and elasticity in adult women. Sci Rep. 2019 Jun 11;9(1):8515. doi: 10.1038/s41598-019-44837-5. PMID 31186509
- [Result] Kuo WH, Jian DW, Wang TG, Wang YC. Neck muscle stiffness quantified by sonoelastography is correlated with body mass index and chronic neck pain symptoms. Ultrasound Med Biol. 2013 Aug;39(8):1356-61. doi: 10.1016/j.ultrasmedbio.2012.11.015. Epub 2013 May 15. PMID 23683408
- [Result] Faria A, Gabriel R, Abrantes J, Bras R, Moreira H. Triceps-surae musculotendinous stiffness: relative differences between obese and non-obese postmenopausal women. Clin Biomech (Bristol). 2009 Dec;24(10):866-71. doi: 10.1016/j.clinbiomech.2009.07.015. Epub 2009 Aug 22. PMID 19703726